CLINICAL TRIAL: NCT03056521
Title: Effect of Preoperative Information About Pain on Postoperative Pain Experience and Patient Satisfaction in Adult Elective Orthopedic Patients: A Randomized Controlled Trial
Brief Title: Effect of Preoperative Information About Pain on Postoperative Pain Experience and Patient Satisfaction
Acronym: epps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/HD07/939U
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The participants and the healthcare providers do not know which patient belongs to which arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Info (Experimental): In this arm the patients are counseled preoperatively about post operative pain.
  Specific information about post operative pain which includes both pharmacologic and non-pharmacologic treatments, complications of pain and benefits of good pain management. This is in addition to the routine care provided
  Interventions: Other: preoperative information about pain
- No info (No Intervention): These patients are in the control group. They are left to receive only the routine preoperative care as made available to them while on ward.

INTERVENTIONS:
Other: preoperative information about pain — It is information about analgesics, post operative pain, complications of pain, benefits of pain treatment and non pharmacologic treatment options.
  Arms: Info

SUMMARY:
Patients are randomized into 2 groups. The intervention group which receives preoperative counseling about pain and a control group which does not receive this counseling.

The patients are followed up looking at pain scores and pain experience and satisfaction with pain management for 2 days post operative.

DETAILED DESCRIPTION:
* All patients admitted for elective upper and lower limb surgery, will be expected to have a preoperative visit by the anesthetic provider on the day before surgery.
* Those who will have consented to participate in the study will be randomized to either the intervention or control group.
* The intervention group will receive specific preoperative information about pain in private by the principal investigator in addition to the preoperative assessment.
* The following variables will be recorded preoperatively: socio-demographics (age, gender, tribe, education level) and vital signs (pulse rate, blood pressure and oxygen saturation).
* A Numerical pain score will be explained to patient before it is recorded preoperatively.
* The patient will also be informed that the pain scores will be repeated after surgery at (someone will take the pain scores again after surgery at) 0, 6, 12, 24, 48hours or till discharge if less than 48hours. In addition the pulse rate, number of analgesic intravenous/ intramuscular injections or tablets needed/or given will be recorded.
* Assessed pain will be classified as no pain (1-3), pain (4-10) but also as no pain (0), mild (1-3), moderate (4-6) and severe pain (7-10).
* Intra operatively, the anaesthetic technique (general or regional), medications given, duration of surgery will be recorded in) the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years and above
* Elective orthopedic surgery patients admitted to orthopedic/trauma ward Mulago hospital
* Patient who gives consent

Exclusion Criteria:

* Patients with chronic pain not related to the surgery they are to undergo
* Patients with bone cancer
* Inability to speak or hear (deaf or dumb)
* Previously recruited but comes for re-surgery for same condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Post operative pain experience (yes or no answer) | 2 days
  Patients subjectively tell you if their pain has been adequately controlled with a yes or no answer
Patient satisfaction (answer yes or no) | 2 days
  Is the patient happy with how the pain has been managed answer yes or no

SECONDARY OUTCOMES:
Time to ambulation | 3 days
  when does the patient start doing some activity with the operated limb less than or greater than 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Moses Othin, Principal Investigator — Makerere University College of Health Sciences
Locations (1):
- Mulago National Referral Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided